CLINICAL TRIAL: NCT06220435
Title: Real-time Image-guided Ultra-hypofractionated Focal Boost to Intraprostatic Lesion(s) With Lymph Node Irradiation for a Very High High-risk Localized Prostate Cancer (the HYPO-RT-PC Boost Trial)
Brief Title: Tumor-directed Radiation Therapy for Patients With the Highest Risk Category of Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPO-RT-PC boost
Record Dates: First submitted 2024-01-10; First posted 2024-01-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: very high risk prostate cancer; radiotherapy; localized prostate cancer treatment; ultra-hypofractionated radiation boost
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYPO-RT-PC boost (Experimental): Ultra-hypofractionated seven-fraction radiotherapy regimen including focal boost and lymph node irradiation.
  Interventions: Radiation: Ultra-hypofractionated radiotherapy regimen.

INTERVENTIONS:
Radiation: Ultra-hypofractionated radiotherapy regimen. — * Prostate tumor(s): 49 Gray (Gy)/7 fractions
  * Prostate gland: 42.7 Gy/7 fractions
  * Elective lymph nodes: 29.4 Gy/7 fractions
  * Seminal vesicles: 31.15 Gy/7 fractions

SUMMARY:
HYPO-RT-PC boost is is an open-label, multicentre, phase II trial evaluating safety and efficacy of real-time image-guided tumor-directed ultra-hypofractionated radiation boost and lymph node irradiation for patients with node-negative high risk localized prostate cancer.

DETAILED DESCRIPTION:
HYPO-RT-PC boost is is an open-label, multicentre, phase II trial evaluating safety and efficacy of real-time image-guided tumor-directed ultra-hypofractionated radiation boost and lymph node irradiation for patients with node-negative high risk localized prostate cancer. 76 participants will be enrolled in the study.

Specific aims of the study are:

* To study the feasibility of ultra-hypofractionation target lesion boost for node-negative very high-risk prostate cancer together with lymph node irradiation (primary outcome).
* To study the effectiveness of ultra-hypofractionated target lesion boost for high-risk prostate cancer.
* To study the feasibility of defining focal boost during concomitant androgen deprivation therapy with advanced functional imaging methods.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >5 years
* Age ≥18 years
* World Health Organization (WHO) performance status 0-2
* Histological evidence of prostate cancer
* Classified as very high-risk according to national guidelines (2-3 of following high risk criteria: T3 / Gleason grade 8 /Prostate-specific antigen (PSA) 20-49 μg/L or and/or Gleason score 9-10 and/or PSA ≥40 μg/L
* At least one Prostate Imaging-Reporting and Data System (PI-RADS) 4-5 lesion on diagnostic Magnetic resonance imaging (MRI)
* Patients must be able to comply with the protocol
* Signed informed consent
* Adequate laboratory findings: haemoglobin (Hb) >90 g/L, absolute neutrophil count >1.0x10^9/l, platelets >75x10^9/l, bilirubin <2.0 x upper limit of normal (ULN), alanine aminotransferase (ALAT) <5x ULN and creatinine <2.0x ULN)

Exclusion Criteria:

* Regional or distant metastasis
* Any contraindications for MRI
* PSA >150 ng/ml
* Previous pelvic radiotherapy
* Prior prostate surgery including transurethral resection of the prostate (TURP)
* Endocrine treatment (past or present)
* Other malignancies than prostate cancer and basalioma in the past five years
* Serious disease state that makes study inclusion and treatment unsuitable
* Severe lower urinary tract symptoms (International Prostate Symptom Score (IPSS) ≥20)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Grade 3+ Genitourinary Adverse Events | start of treatment - 5 years
  Acute grade 3+ genitourinary Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Grade 2+ Genitourinary Adverse Events | start of treatment - 5 years
  Acute grade 2+ genitourinary Adverse Events according to CTCAE v5.0.
Failure-free survival | consent date - 5 years
Local failure-free survival | enrollment date - 5 years
Biochemical failure-free survival | enrollment date - 5 years
Cancer-specific survival | enrollment date - 5 years
Overall survival failure-free survival, cancer-specific survival, and overall survival | enrollment date - 5 years
Distant metastasis-free survival failure-free survival, cancer-specific survival, and overall survival | enrollment date - 5 years
Time to systemic therapy failure-free survival, cancer-specific survival, and overall survival | enrollment date - 5 years
Adverse Events according to CTCAE v5.0 | start of treatment - 5 years
Health-related quality of life assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C-30) | inclusion date - 5 years
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
Health-related quality of life assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire PR-25 (EORTC QLQ-PR25) | inclusion date - 5 years
  It includes subscales assessing urinary symptoms, bowel symptom), treatment-related symptom) and sexual functioning with score from 0 to 4 per item. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Adalsteinn Gunnlaugsson, MD, PhD, Principal Investigator — Region Skåne, Lund University
Locations (2):
- Sweden (2):
  - Region Skåne, Skåne University Hospital, Lund
  - Region Västerbotten, Umeå University Hospital, Umeå

IPD SHARING:
Plan to Share IPD: No